CLINICAL TRIAL: NCT00982423
Title: To Define the Effects of Decreasing the Furosemide Dose on Cardiorenal and Humoral Function in Humans With Compensated Chronic Heart Failure (CHF) With and Without Renal Dysfunction
Brief Title: The Effects of Decreasing the Lasix Dose on the Cardiorenal System
Acronym: Aim1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Horng Chen, MD, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-003210; R01HL084155 (NIH); P01HL076611 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2009-09-18; First posted 2009-09-23 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure; Kidney Dysfunction
Keywords: heart failure; heart failure with and without kidney dysfunction
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Furosemide (Experimental): Subjects received their clinically prescribed dose of furosemide for a 3 week stabilization period, then were assessed for cardiorenal and humoral function. Subjects then had a 50% reduction of the furosemide dose for a 3 week stabilization period, and were assessed for cardiorenal and humoral function again.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Subjects received their clinically prescribed dose of furosemide for a 3 week stabilization period, then were assessed for cardiorenal and humoral function. Subjects then had a 50% reduction of the furosemide dose for a 3 week stabilization period, and were assessed for cardiorenal and humoral function again.
  Other Names: Lasix

SUMMARY:
The investigators' objective is to define the effects of decreasing the furosemide dose on heart, kidney and humoral function in people with compensated heart failure and kidney dysfunction and also in people with compensated heart failure without kidney dysfunction. Secondly, to define the humoral activation in both groups.

DETAILED DESCRIPTION:
The broad objective of this protocol is to advance our understanding of the pathophysiological mechanisms of human Cardiorenal Syndrome (CRS) with a specific emphasis upon the biological interaction between diuretic therapy, the renin-angiotensin-aldosterone-system (RAAS) and cyclic 3'-5'-guanosine monophosphate (cGMP) pathway.

ELIGIBILITY:
Inclusion Criteria for Subjects with Compensated CHF without Renal Dysfunction:

* Left ventricular ejection fraction of equal or less than 40% assessed by echocardiography, nuclear scan, MRI, or left ventriculogram within the past 36 months.
* Stable New York Heart Association (NYHA) class II and III symptoms as defined by: a) no change in NYHA symptoms over the past 3 months; b) on stable doses of ACE inhibitor or beta blocker or digoxin or furosemide or angiotensin II receptor, type 1 (AT1) blocker over the past 3 months; c) no episode of decompensated CHF over the past 6 months.
* Calculated creatinine clearance of equal or less than 80 ml/min, using the Cockcroft-Gault formula assessed within the past 36 months and a confirmatory calculated creatinine clearance equal or less than 80 ml/min at the time of enrollment.

Inclusion Criteria for Subjects with Compensated CHF with Renal Dysfunction:

* Left ventricular ejection fraction of equal or less than 40% assessed by echocardiography, nuclear scan or left ventriculogram within the past 36 months.
* Stable New York Heart Association (NYHA) class II and III symptoms as defined by: a) no change in NYHA symptoms over the past 3 months; b) on stable doses of ACE inhibitor or beta blocker or digoxin or furosemide or AT1 blocker over the past 3 months; c) no episode of decompensated CHF over the past 6 months.
* Calculated creatinine clearance of equal or less than 60 ml/min and greater than 20 ml/min, using the Cockcroft-Gault formula assessed within the past 36 months and a confirmatory calculated creatinine clearance equal or less than 60 ml/min and greater than 20 ml/min at the time of enrollment.

Exclusion Criteria for both groups:

* Prior diagnosis of intrinsic renal diseases including renal artery stenosis of > 50%
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Patients who are taking aldosterone antagonist
* Hospitalization for decompensated CHF during the past 6 months
* Subjects on other diuretics besides furosemide
* Myocardial infarction within 6 months of screening
* Unstable angina within 6 months of screening or any evidence of myocardial ischemia
* Significant valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening or other evidence of significantly compromised central nervous system (CNS) perfusion
* Alanine Aminotransferase (ALT) result >1.5 times the upper limit of normal
* Serum sodium of < 125 milliequivalent (mEq)/dL or > 150 mEq/dL
* Serum potassium of < 3.5 mEq/dL or > 5.5 mEq/dL
* Serum digoxin level of > 2.0 ng/ml
* Hemoglobin < 10 gm/dl
* Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* Received an investigational drug within 1 month prior to dosing
* Patients with an allergy to iodine.
* Female subject who is pregnant or breastfeeding
* In the opinion of the investigator is unlikely to comply with the study protocol or is unsuitable for any reason.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H Chen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] McKie PM, Schirger JA, Benike SL, Harstad LK, Chen HH. The effects of dose reduction of furosemide on glomerular filtration rate in stable systolic heart failure. JACC Heart Fail. 2014 Dec;2(6):675-7. doi: 10.1016/j.jchf.2014.05.014. Epub 2014 Sep 24. No abstract available. PMID 25262369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from outpatients being treated at the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: There was 1 screen failure and 8 subjects withdrew prior to group assignment: 1 due to chest pain, 1 due to surgical procedure scheduled to take place during treatment phase, 1 due to fluid overload, 2 due to time constraints of work and family issues, and 3 due to primary physician-initiated medication titration.
Groups:
- Compensated CHF Without Renal Dysfunction: Preserved renal function was defined as glomerular filtration rate (GFR) greater than or equal to 60 mg/min/1.73m^2.
- Compensated CHF With Renal Dysfunction: Renal Dysfunction was defined as GFR less than 60 mg/min/1.73m^2.
Period: Overall Study
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Started | 13 | 19
Completed | 13 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Compensated CHF Without Renal Dysfunction: Preserved renal function was defined as GFR greater than or equal to 60 mg/min/1.73m^2.
- Total: Total of all reporting groups
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction | Total
Number analyzed (Participants) | 13 | 19 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (3) | 76 (2) | 72.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 9 | 13 | 22
Region of Enrollment [Number; unit: participants]
  United States | 13 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Renal Function as Measured by Glomerular Filtration Rate (GFR) at Baseline and in Response to Decreasing Furosemide Dose
Description: Kidney function was measured by GFR determined by iothalamate clearance. GFR describes the flow rate of filtered fluid through the kidney measured in milliliters per minute per 1.73 m^2 of body surface area. A lower GFR means the kidney is not filtering normally. An estimated GFR of less than 60 mg/min/1.73 m^2 of body surface area is considered to be impaired kidney function.
Time Frame: 3 weeks, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Number analyzed (Participants) | 13 | 19
ml/min
  Baseline (3 weeks) | 77 (3) | 42 (3)
  Approximately 6 weeks | 73 (5) | 50 (4)
Statistical Analysis 1: Comparison: Compensated CHF With Renal Dysfunction; Comparison between baseline dose of furosemide (3 weeks) versus reduced dose of furosemide (approximately 6 weeks); Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Compensated CHF With Renal Dysfunction; Comparison between GFR taken at baseline dose Furosemide (3 weeks) versus normal GFR; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Renal Plasma Flow at Baseline and in Response to Decreasing Furosemide Dose
Description: Effective renal plasma flow (eRPF) is a measure used to calculate renal plasma flow (RPF) and hence estimate renal function. Renal plasma flow is the volume of blood plasma that flows through the kidneys per unit time, measured as ml/min.
Time Frame: 3 weeks, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Number analyzed (Participants) | 13 | 19
ml/min
  Baseline (3 weeks) | 304 (19) | 198 (20)
  Approximately 6 weeks | 293 (23) | 214 (21)

3. Secondary Outcome: Aldosterone at Baseline and in Response to Decreasing Furosemide Dose
Description: Aldosterone is part of the renin-angiotensin-aldosterone system (RAAS). Drugs that interfere with the secretion or action of aldosterone are in use as antihypertensives, like lisinopril, which lowers blood pressure by blocking the angiotensin-converting enzyme (ACE), leading to lower aldosterone secretion. The net effect of these drugs is to reduce sodium and water retention but increase retention of potassium.
Time Frame: 3 weeks, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Number analyzed (Participants) | 13 | 19
ng/dL
  Baseline (3 weeks) | 7.9 (1.8) | 4.9 (0.6)
  Approximately 6 weeks | 7.6 (1.3) | 4.9 (0.6)

4. Secondary Outcome: Plasma Renin Activity at Baseline and in Response to Decreasing Furosemide Dose
Description: Plasma renin activity is a measure of the activity of the plasma enzyme renin, which plays a major role in the body's regulation of blood pressure, thirst, and urine output. Renin is an enzyme that hydrolyses angiotensinogen secreted from the liver into the peptide angiotensin I. Renin's primary function is to cause an increase in blood pressure, leading to restoration of perfusion pressure in the kidneys.
Time Frame: 3 weeks, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Number analyzed (Participants) | 13 | 19
ng/mL/hr
  Baseline (3 weeks) | 4.3 (2.0) | 2.1 (0.8)
  Approximately 6 weeks | 2.7 (1.1) | 1.4 (0.5)

5. Secondary Outcome: Angiotensin II at Baseline and in Response to Decreasing Furosemide Dose
Description: Renin activates the renin-angiotensin system by cleaving angiotensinogen, produced by the liver, to yield angiotensin I, which is further converted into angiotensin II by the angiotensin-converting enzyme (ACE) primarily within the capillaries of the lungs. Angiotensin II then constricts blood vessels, increases the secretion of antidiuretic hormone (ADH) and aldosterone, and stimulates the hypothalamus to activate the thirst reflex, each leading to an increase in blood pressure.
Time Frame: 3 weeks, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Number analyzed (Participants) | 13 | 19
pg/mL
  Baseline (3 weeks) | 3.3 (0.6) | 3.1 (0.7)
  Approximately 6 weeks | 3.4 (1.0) | 3.2 (0.9)

6. Secondary Outcome: Plasma Cyclic Guanosine Monophosphate (cGMP) at Baseline and in Response to Decreasing Furosemide Dose
Description: Any change in atrial filling pressures leads to the release of atrial natriuretic peptides (ANP) from the heart. Once released, atrial peptides exert potent direct vasodilator and natriuretic actions by virtue of the ability to increase their intracellular second messenger, cGMP. Plasma cGMP correlates closely with the severity of congestive heart failure.
Time Frame: 3 weeks, approximately 6 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Number analyzed (Participants) | 13 | 19
pg/mL
  Baseline (3 weeks) | 5.0 (0.9) | 5.7 (0.8)
  Approximately 6 weeks | 4.6 (0.7) | 7.0 (1.0)
Statistical Analysis 1: Comparison: Compensated CHF With Renal Dysfunction; Comparison between reduced dose Furosemide and baseline dose Furosemide; Test type: Superiority or Other; p = 0.075, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Subjects received weekly phone calls from the study coordinator to address any concerns and to collect safety information.
Arm/Group | Compensated CHF Without Renal Dysfunction | Compensated CHF With Renal Dysfunction
Serious Adverse Events (participants affected / at risk) | 0/13 | 2/19
Other Adverse Events (participants affected / at risk) | 0/13 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compensated CHF Without Renal Dysfunction (N=13) | Compensated CHF With Renal Dysfunction (N=19)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compensated CHF Without Renal Dysfunction (N=13) | Compensated CHF With Renal Dysfunction (N=19)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes